CLINICAL TRIAL: NCT05821920
Title: Prospective Multicentric Clinical Study to Assess Safety of MUST MINI Posterior Cervical System.
Brief Title: A Safety Study on Posterior Pedicle Screw System
Acronym: MUST MINI PMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P05.008.01
Record Dates: First submitted 2023-04-04; First posted 2023-04-20 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2023-04

CONDITIONS: Degenerative Disc Disease; Trauma Injury; Tumor
MeSH Terms: conditions — Intervertebral Disc Degeneration; Accidental Injuries; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: MUST MINI system — cervical posterior fixation system

SUMMARY:
The goal of this study is to assess the MUST MINI system safety in patient who will undergo a posterior cervical spine fusion intervention. Patients will be invited to partecipate during preoperative visit and follow the postoperative visits according to the standard practice.

DETAILED DESCRIPTION:
Patient who will undergo a posterior cervical spine fusion intervention, will be invited during preoperative visit to take part to the study.

The study is an observational multicentric study with an enrolment period of 12 months with the aim to assess the safety of MUST MINI system.

All adverse events will be collected for all study duration, classified as device and not device related. Screw failure rate is calculated considering screw loosening, breakage, lost-reduction events.

Standard radiological investigations are previewed at preoperative visit, before discharge and at 6 weeks and 12 months follow-up after surgery visits; the risk of any further exposure to radiation other than it's routine use in a diagnostic manner within the follow-up period can be excluded.

A final visit at 12 months level index fusion will be evaluated clinically as well as radiographically, with a confirmation CT scan as per standard of care. Screw placement accuracy will be evaluated during this visit.

A functional cervical x-ray is considered also during last follow-up (12 months after surgery) in order to assess cervical spine functionality.

ELIGIBILITY:
Inclusion Criteria:

* those affected by degenerative disc disease needing a posterior surgical instrumented treatment aimed at segmental fusion,
* those who will undergo posterior fixation due to traumatic lesion or tumor,
* Patients with BMI ≤ 35 kg/m2,
* those who signed the consent form to participate to the study.

Exclusion Criteria:

* Patients <18 years,
* Patients who are pregnant or intend to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will undergo a posterior cervical spine fusion with MUST MINI system and respecting the inclusion criteria will be invited to participate to the study during the preoperative visit
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of MUST MINI system safety | 24 months
  collection of adverse event

SECONDARY OUTCOMES:
Clinical outcomes | preop, 6 weeks, 6 months, 12 months
  mJOA questionnaire, a 18-point investigator-administered scale separately addresses motor dysfunction of the upper extremity (MDUE) and motor dysfunction of the lower extremity (MDLE), sensory loss of the upper extremity, and sphincter dysfunction (SD). Severe myelopathy (0-11), moderate myelopathy (12-14), mild myelopahty (15-17).
Clinical outcomes | preop, 6 weeks, 6 months, 12 months
  NDI questionnaire. Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
  0-4points (0-8%) no disability, 5-14points ( 10 - 28%) mild disability, 15-24points (30-48% ) moderate disability, 25-34points (50- 64%) severe disability, 35-50points (70-100%) complete disability
Clinical outcomes | preop, 6 weeks, 6 months, 12 months
  EQ-5D questionnaire consists of two section, descriptive and a visual analog scale to describe the own health status. The score is calculated by assigning a numerical value to each response level (i.e., 1 for "no problems", 5 for "extreme problems"/"unable to") and summing these values across the five items, resulting in a score from 5 to 25.
Clinical outcomes | preop, 6 weeks, 6 months, 12 months
  VAS pain scale measure the pain intensity with a scale from 0 ('no pain') to 10 ('pain as bad as it could possibly be').
Bone fusion at index level | 12 month
  For each level a CT examination will be performed in order to define if bone fusion is or not. The presence or absence of bridging trabecular bone across the segment can identify is reported.
Cervical spine functionality | Immediate postop, 6 weeks, 12 months
  Sandard functional x-ray is performed in order to measure the segmental range of motion in the lumbar spine during flexion-extension with the purpose of gathering additional data for the diagnosis of instability.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Lehmberg, Prof Med, Principal Investigator — München Klinik Bogenhausen
Locations (1):
- München Klinik Bogenhausen, München, Germany

IPD SHARING:
Plan to Share IPD: No